CLINICAL TRIAL: NCT00828308
Title: BrUOG-PROS-221 Neoadjuvant Weekly Ixabepilone for High Risk, Clinically Localized Prostate Cancer: A Phase II Study
Brief Title: Neoadjuvant Weekly Ixabepilone for High Risk, Clinically Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG-Pros-221
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
Keywords: localized; high risk; prostate cancer; neoadjuvant treatment
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ixabepilone; Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ixabepilone (Experimental): Ixabepilone, 16 mg/m2 or 20mg/m2, weekly x 3, in 4 week cycles, x 4 cycles.
  Prostatectomy 2-8 weeks after completion ***this was standard of care and not a part of the study***
  Interventions: Drug: Ixabepilone; Procedure: Prostatectomy

INTERVENTIONS:
Drug: Ixabepilone — Ixabepilone, 16 mg/m2 or 20mg/m2, weekly x 3, in 4 week cycles, x 4 cycles.
  Other Names: Ixempra
Procedure: Prostatectomy — Prostatectomy 2-8 weeks after completion ***this was standard of care and not a part of the study**
  Other Names: Prostatectomy 2-8 weeks after completion ***this was standard of care and not a part of the study**

SUMMARY:
Ixabepilone, 16 mg/m2 or 20mg/m2, weekly x 3, in 4 week cycles, x 4 cycles.

Prostatectomy 2-8 weeks after completion(standard of care and not a part of study)

DETAILED DESCRIPTION:
Ixabepilone, 16 mg/m2 or 20mg/m2, weekly x 3, in 4 week cycles, x 4 cycles. Prostatectomy 2-8 weeks after completion of chemotherapy (this was standard of care).

This protocol evaluated weekly ixabepilone prior to robotic prostatectomy for patients with high risk localized prostate cancer. PSA response rate, tumor margin status and pathologic responses were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of prostatic adenocarcinoma. Patients with small cell, neuroendocrine or transitional cell carcinomas are not eligible.
* All eligible patients must have a known Gleason sum based on biopsy or TURP at the time of registration.
* Clinically Localized Disease: Patients must have clinical stage T1-T3a and no radiographic evidence of metastatic disease as demonstrated by:
* Either CT or MRI of the abdomen and pelvis, that demonstrate no nodes > 1 cm: or endorectal MRI(If one or more lymph nodes(s) measures > 1 cm, a negative biopsy is required.)
* Negative bone scan (with plain films and /or MRI and/or CT scan confirmation, if necessary).(Positive PET and Prostascint scans are not considered proof of metastatic disease.)
* Patients must have high risk disease defined as either:

  * Gleason Score 8-10
  * PSA > 15 ng/ml
  * Stage T3a
  * Stage T2c and Gleason score of 7
  * Stage T2b, Gleason score of 7, greater than 50% of the cores positive from a single lobe.
* No prior treatment for prostate cancer including prior surgery (excluding TURP), pelvic lymph node dissection, radiation therapy, chemotherapy or hormone therapy.
* Patient must be appropriate candidates for radical prostatectomy with an estimated life expectancy > 10 years as determined by an urologist.
* ECOG PS 0-1
* Age > 18 years of age.
* Required initial laboratory values:

  * ANC > 1500/ul
  * Platelet count > 100,000/mm3
  * Creatinine < 2.0 mg/dl
  * Serum PSA < 100 ng/ml
  * Bilirubin < upper institutional limit of normal (ULN)
  * AST/ALT < 2.5 X ULN

Exclusion Criteria:

* Active or uncontrolled infection.
* Patients must not have other coexistent medical condition that would preclude protocol therapy.
* Previous severe hypersensitivity reaction to a drug formulated in CremophoreL (polyoxyethylated castor oil).
* Grade 1 or greater neuropathy (motor or sensory) at study entry

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Study Chair — BrUOG Study Chair
Locations (1):
- Miriam Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled 2/11/09 and last patient enrolled was 3/30/11
Groups:
- Ixabepilone: Ixabepilone, 16 mg/m2 or 20mg/m2, weekly x 3, in 4 week cycles, x 4 cycles. Prostatectomy 2-8 weeks after completion of chemotherapy.
Period: Overall Study
Arm/Group | Ixabepilone
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ixabepilone: Ixabepilone, 16 mg/m2, weekly x 3, in 4 week cycles, x 4 cycles. Prostatectomy 2-8 weeks after completion of chemotherapy (this was standard of care and not a part of the study)
Arm/Group | Ixabepilone
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Prostate-Specific Antigen (PSA) Response
Description: Decrease in PSA:number of participants with decreased serum PSA level after 12 weeks of ixabepilone
Time Frame: after 12 weeks of ixabepilone
Measure: Number; unit: participants
Groups:
- Ixabepilone: Ixabepilone, 16 mg/m2 or 20mg/m2, weekly x 3, in 4 week cycles, x 4 cycles. Prostatectomy will occur 2-8 weeks after completion of chemotherapy.
Arm/Group | Ixabepilone
Number analyzed (Participants) | 16
participants | 14

ADVERSE EVENTS:
Time Frame: Toxicities collected during treatment and approximately 30 days post last dose of drug (approximately 5 months). Of note, the adverse events posted are all AEs patient's experienced and do not equate to toxicities confirmed as related to treatment.
Arm/Group | Ixabepilone
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixabepilone (N=16)
pneumonia (3) with normal ANC, post infuection bronchitis (3), wheezing (3) (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixabepilone (N=16)
Constipation (Investigations) | 6 (6)
nasuea (Investigations) | 3 (3)
neuorapthy (Investigations) | 13 (13)
fatigue (Investigations) | 11 (11)
diarrhea (Investigations) | 7 (7)
taste alteration (Investigations) | 3 (3)
heartburn (Investigations) | 1 (1)
pain (Investigations) | 1 (1)
dehydration (Investigations) | 3 (3)
insomnia (Investigations) | 4 (4)
wt loss (Investigations) | 3 (3)
rash/pruritus (Investigations) | 2 (2)
anorexia (Investigations) | 1 (1)
hyperpigmentation (Investigations) | 1 (1)
abdominal cramping/pain (Investigations) | 4 (4)
dysphagia (Investigations) | 1 (1)
urinary frequency (Investigations) | 2 (2)
allergic reaction/hypersensitivity reaction (Investigations) | 3 (3)
edema (Investigations) | 1 (1)
rhinitis (Investigations) | 2 (2)
depression (Investigations) | 1 (1)
infection (Investigations) | 4 (4)
alopecia (Investigations) | 5 (5)
HTN (Investigations) | 1 (1)
shortness of breath (Investigations) | 1 (1)
headache (Investigations) | 1 (1)
muscle aches/myalgia (Investigations) | 2 (2)
wheezing (Investigations) | 1 (1)
cough (Investigations) | 1 (1)
WBC (Investigations) | 1 (1)
ANC (Investigations) | 1 (1)
HGB (Investigations) | 2 (2)
pain-joint (Investigations) | 1 (1)
sore throat (Investigations) | 3 (3)
flushing (Investigations) | 1 (1)
flatulence (Investigations) | 1 (1)
mood (Investigations) | 1 (1)
pain-mouth (Investigations) | 1 (1)
pain-muscle (Investigations) | 1 (1)
hoarseness (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No